CLINICAL TRIAL: NCT00245921
Title: A Phase 3, Multicenter, Open-Label Study to Evaluate the Safety and Efficacy of Levonorgestrel 90 mg and Ethinyl Estradiol 20 mg in a Continuous Daily Regimen for Oral Contraception
Brief Title: Study Evaluating Levonorgestrel and Ethinyl Estradiol for Oral Contraception
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 0858A2-313, 314, 320; B3211019, B3211020, B3211022 (Other: Pfizer)
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2006-05

CONDITIONS: Contraception
Keywords: contraception
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol

INTERVENTIONS:
Drug: Levonorgestrel 90 mg/Ethinyl Estradiol 20 mg

SUMMARY:
To evaluate the safety and contraceptive efficacy of an oral contraceptive containing a combination of LNG 90 mg/EE 20 mg in a continuous-use regimen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18 to 49 years
* Regular (21- to 35- day) menstrual cycles for the 3-month period preceding visit 1
* Must be sexually active and at risk for becoming pregnant.

Exclusion Criteria:

* Planned use of any other form of birth control other than the test article.
* Depression requiring hospitalization or associated with suicidal ideation within the last 3 years.
* High blood pressure (defined as elevated sitting blood pressure: > 140/90 mm Hg).

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2000
Dates: Start 2003-02; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and contraceptive efficacy

SECONDARY OUTCOMES:
To evaluate the effects of this LNG/EE combination on bleeding profile, endometrial histology, hemostasis measures, hemoglobin levels, discontinuation rates, subject satisfaction, and cycle-related symptoms and work productivity at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Reid RL, Fortier MP, Smith L, Mirkin S, Grubb GS, Constantine GD. Safety and bleeding profile of continuous levonorgestrel 90 mcg/ethinyl estradiol 20 mcg based on 2 years of clinical trial data in Canada. Contraception. 2010 Dec;82(6):497-502. doi: 10.1016/j.contraception.2010.06.002. Epub 2010 Jul 16. PMID 21074011